CLINICAL TRIAL: NCT04532463
Title: Clinical Effectiveness and Safety of Amphotericin B With Flucytosine-Fluconazole Therapy for Cryptococcal Meningitis in Patients With HIV Infection
Brief Title: Clinical Effectiveness and Safety of Amphotericin B With Flucytosine-Fluconazole Therapy for Cryptococcal Meningitis
Status: Completed | Type: Observational
Sponsor: University of Pharmacy, Yangon (Other)
Responsible Party: Principal Investigator, Ms. Zin Win May, Principal Investigator, Clinical effectiveness and safety of Amphotericin B with Flucytosine-Fluconazole therapy for Cryptococcal meningitis in patients with HIV infection, University of Pharmacy, Yangon
Other Study IDs: 122020
Record Dates: First submitted 2020-08-18; First posted 2020-08-31 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Cryptococcal Meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — Amphotericin B; Flucytosine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Amphotericin B,Flucytosine, Fluconazole: Amphotericin B 1 mg/kg 1 week & Flucytosine 100 mg/kg 1 week followed by Fluconazole 1200 mg/day 1 week
  Interventions: Drug: Amphotericin B 1 mg/kg 1 week & Flucytosine 100 mg/kg 1 week followed by Fluconazole 1200 mg/day 1 week

INTERVENTIONS:
Drug: Amphotericin B 1 mg/kg 1 week & Flucytosine 100 mg/kg 1 week followed by Fluconazole 1200 mg/day 1 week — To study the clinical effectiveness and safety of amphotericin B with flucytosine-fluconazole therapy for cryptococcal meningitis in patients with HIV infection.

SUMMARY:
To study the clinical effectiveness and safety of amphotericin B with flucytosine-fluconazole therapy for cryptococcal meningitis in patients with HIV infection.

DETAILED DESCRIPTION:
Cryptococcal meningitis is an AIDS-defining illness mostly caused by the fungus, Cryptococcus neoformans. In high-income countries, the use of amphotericin B in combination with a more expensive drug, flucytosine, is most effective for the management of cryptococcal meningitis; but access to flucytosine is severely limited in middle and low-income countries. In Myanmar, currently recommended regimen for cryptococcal meningitis are combination of amphotericin B with fluconazole. Although amphotericin plus flucytosine followed by fluconazole therapy is the currently preferred regimen in WHO treatment guidelines, it is not still commonly used in Myanmar clinical practice because of its limited availability. Therefore, the data regarding tolerability and clinical effectiveness of flucytosine are unavailable for Myanmar patients.

Although trials were carried out for investigating the effectiveness of flucytosine in the HIV population of Africa, the variability in drug response can occur in Myanmar patients due to the racial and genetic differences and whether it is effective and safe for Myanmar people is a great curiosity question for clinicians and healthcare workers. In Myanmar, amphotericin plus flucytosine followed by fluconazole regimen will be supplied by National AIDS Program (NAP) and indicated in 2020. Thus, the documents for effectiveness and safety profile need to be established. This is the reason that the effectiveness and safety of amphotericin B with flucytosine and fluconazole combination therapy should be studied. From this study, it can provide information to physicians regarding the effectiveness as well as safety of those drugs in the management of cryptococcal meningitis in HIV patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HIV-associated cryptococcal meningitis, admitted to inpatient department of SHW, SHM, SHT, YGH, NOGTH and IGH during the study period
2. Patients of both sexes
3. Age above 14 years
4. Patients or caregivers who will give informed consent to participate in this study

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to SHW, SHM, SHT, YGH, NOGTH and IGH with HIV-associated cryptococcal meningitis who will be treated with amphotericin + flucytosine + fluconazole induction regimen.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Clinical effectiveness | 14 days (day1 to day 14)
  1. To describe the clinical effectiveness of amphotericin B with flucytosine-fluconazole combination therapy by assessing clinical parameters (presence of headache, fever, convulsion, abnormal mental status and death) at day 1, day 7 and day 14
  2. To determine the severity of headache before and after treatment by numerical rating scale
Clinical safety | 14 days (day1 to day 14)
  3. . To describe the clinical safety of amphotericin B with flucytosine-fluconazole combination therapy by assessing hematological and biochemical parameters (hemoglobin, neutrophil, platelet, ALT, AST, serum creatinine and serum potassium level ) by DAIDS grading at baseline, day 7 and day 14

SECONDARY OUTCOMES:
back-ground characteristics of patients | 14 days (day1 to day 14)
  4. To find out the back-ground characteristics of patients (age,gender) with HIV-associated cryptococcal meningitis

CONTACTS AND LOCATIONS:
Overall Officials: zin win may, B.Pharm, Principal Investigator — Specialist Hospital Thakeyta
Locations (1):
- Specialist hospital Mingalardon,Thakeyta and Waibargi,Yangon General Hospital,Insein General Hospital, North Oakalapa General and Teaching Hosptial, Yangon, Burma

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT04532463/Prot_SAP_ICF_000.pdf